CLINICAL TRIAL: NCT03336970
Title: Efficacy of Chlorhexidine as a Final Irrigant in Single-visit Root Canal Treatment: A Prospective Comparative Study
Brief Title: Efficacy of Chlorhexidine as a Final Irrigant in Single-visit Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Kemal Çalışkan (Other)
Responsible Party: Sponsor-Investigator, Mehmet Kemal Çalışkan, Prof.Dr., Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Single visit study
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Root Canal Infection
Keywords: single visit root canal treatment, chlorhexidine
MeSH Terms: interventions — Edetic Acid; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single visit root canal treatment (Active Comparator): The teeth were treated in single-visit (SV) root canal treatment. Final root canal irrigation was performed with 5% EDTA, followed by 2.5% NaOCl and received an additional final rinse with 2% CHX before obturation.
  Interventions: Other: EDTA; Other: NaOCl; Other: CHX
- Multiple visit root canal treatment (Active Comparator): The teeth were treated in multiple visit (MV) root canal treatment. After completion of root canal instrumentation, calcium hydroxide paste was placed into the root canal. In second visit, all root canals were irrigated with 5% EDTA followed by 2.5% NaOCl before obturation.
  Interventions: Other: EDTA; Other: NaOCl; Other: Calcium hydroxide

INTERVENTIONS:
Other: EDTA
Other: NaOCl
Other: CHX
  Arms: Single visit root canal treatment
Other: Calcium hydroxide
  Arms: Multiple visit root canal treatment

SUMMARY:
Ninety asymptomatic maxillary anterior teeth with periapical lesions were treated in single versus multiple visit root canal treatment. Half of the teeth were randomly assigned to the single-visit (SV) group and received an additional final rinse with 2% CHX before obturation. The other teeth were treated in multiple visits (MV) with calcium hydroxide dressing. All patients were recalled and investigated clinically and radiographically for 24 months.

DETAILED DESCRIPTION:
The aim of the study was to evaluate postoperative pain and radiographic evidence of periapical healing in teeth with apical periodontitis treated in a single visit with an additional final irrigation using 2% chlorhexidine and to compare the results with conventional multiple-visit root canal treatment (RCT) with an intracanal calcium hydroxide dressing as a control group. Ninety asymptomatic maxillary anterior teeth with periapical lesions were treated by a single operator using the step-back technique with manual instrumentation with 2.5% sodium hypochlorite (NaOCl) and 5% ethylenediaminetetraacetic acid (EDTA) as irrigants. Half of the teeth were randomly assigned to the single-visit (SV) group and received an additional final rinse with 2% chlorhexidine (CHX) before obturation. The other teeth were treated in multiple visits (MV), after completion of root canal instrumentation calcium hydroxide paste was placed into the root canal and root canal obturation was performed in second visit. All patients were recalled and investigated clinically and radiographically for 24 months. Postoperative pain at 24-48 hours and changes in apical bone density indicating radiographic healing were evaluated statistically using the Mann-Whitney U-test followed by the Friedman and the Wilcoxon tests (α=.05).

ELIGIBILITY:
Inclusion Criteria:

* patients with a non-contributory medical history,
* mature maxillary anterior teeth with periapical lesions (< 5 mm),
* diagnosed as asymptomatic apical periodontitis.

Exclusion Criteria:

* clinical symptoms, drainage,
* more than 5 mm loss of periodontal attachment,
* previous endodontic treatment,
* non-restorable tooth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
The rate of radiographic healing of the periapical lesion | 6,12 and 24 months
  Follow-up visits were performed after 6, 12 and 24 months for all patients in order to evaluate radiographic status. Changes in apical bone density indicating radiographic healing was assessed by the periapical index (PAI).

SECONDARY OUTCOMES:
The level of postoperative pain | 24 hours and 48 hours
  Postoperative pain after 24 and 48 hours, was measured using a modified 4-grade visual analogue scale (VAS) ranging from 1 (no pain), 2 (mild pain), 3 (moderate pain/pain relieved by analgesics), to 4 (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Seniha Miçooğulları Kurt, Principal Investigator — Ege University Faculty of Dentistry; Mehmet Kemal Çalışkan, Study Director — Ege University Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729
- [Background] Penesis VA, Fitzgerald PI, Fayad MI, Wenckus CS, BeGole EA, Johnson BR. Outcome of one-visit and two-visit endodontic treatment of necrotic teeth with apical periodontitis: a randomized controlled trial with one-year evaluation. J Endod. 2008 Mar;34(3):251-7. doi: 10.1016/j.joen.2007.12.015. PMID 18291270
- [Background] El Mubarak AH, Abu-bakr NH, Ibrahim YE. Postoperative pain in multiple-visit and single-visit root canal treatment. J Endod. 2010 Jan;36(1):36-9. doi: 10.1016/j.joen.2009.09.003. PMID 20003932
- [Background] Zamany A, Safavi K, Spangberg LS. The effect of chlorhexidine as an endodontic disinfectant. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Nov;96(5):578-81. doi: 10.1016/s1079-2104(03)00168-9. PMID 14600693
- [Background] Peters LB, Wesselink PR. Periapical healing of endodontically treated teeth in one and two visits obturated in the presence or absence of detectable microorganisms. Int Endod J. 2002 Aug;35(8):660-7. doi: 10.1046/j.1365-2591.2002.00541.x. PMID 12196219
- [Background] Rocas IN, Provenzano JC, Neves MA, Siqueira JF Jr. Disinfecting Effects of Rotary Instrumentation with Either 2.5% Sodium Hypochlorite or 2% Chlorhexidine as the Main Irrigant: A Randomized Clinical Study. J Endod. 2016 Jun;42(6):943-7. doi: 10.1016/j.joen.2016.03.019. Epub 2016 Apr 30. PMID 27142579